CLINICAL TRIAL: NCT02176525
Title: Safety, Antiviral Activity, and Pharmacokinetics of Multiple Oral Doses of BI 207127 NA Administered q8H for 5 Days as Monotherapy, a Randomised, Double-blind, Placebo Controlled Study
Brief Title: Multiple Oral Doses of BI 207127 NA in Treatment naïve and Treatment-experienced Hepatitis C Virus (HCV)-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1241.2
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

ARMS (3):
- BI 207127 in patients with cirrhosis (Experimental): multiple rising doses
  Interventions: Drug: BI 207127 NA
- BI 207127 in patients without cirrhosis (Experimental): multiple rising doses
  Interventions: Drug: BI 207127 NA
- Placebo in patients without cirrhosis (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 207127 NA
  Arms: BI 207127 in patients with cirrhosis; BI 207127 in patients without cirrhosis
Drug: Placebo
  Arms: Placebo in patients without cirrhosis

SUMMARY:
The purpose of this study was to investigate antiviral activity, safety and pharmacokinetics of 5 days of monotherapy with BI 207127 in HCV genotype 1 (GT1) infected patients. Both treatment-naïve patients and patients previously treated with peginterferon and ribavirin were included. In addition, the effect of study medication was examined in a group of patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 - 70 years
* Male OR female with documented hysterectomy OR menopausal female with last menstrual period at least 12 months prior to screening
* Written informed consent consistent with International Conference on Harmonization/Good Clinical Practice and local legislation given prior to any study procedures
* Chronic HCV infection demonstrated by positive HCV immunoglobulin G Antibody
* HCV genotype 1 which has to be confirmed by central laboratory test before Visit 2
* For non-cirrhotic cohorts: Liver biopsy obtained within the last 36 months consistent with HCV infection showing minimal to mild liver fibrosis and without cirrhosis (Ishak or Metavir grade ≤ 2). For cirrhotic cohorts, previous liver biopsy or Fibroscan consistent with liver cirrhosis performed at any time before screening
* HCV RNA load > 100,000 IU RNA per ml serum at screening

Exclusion Criteria:

* All fertile males not willing to use an adequate form of contraception (condom, sterilisation at least 6 months post operation) in case their partner is of childbearing potential and is not using an adequate form of contraception (hormonal contraceptives, oral or injectable/ implantable, intra-uterine device)
* Patients who have been treated with at least one dose of any HCV-polymerase inhibitor for acute or chronic hepatitis C infection
* Any other or additional plausible cause for chronic liver disease, including the presence of other viruses known or suspected to cause hepatitis
* Decompensated liver disease within past 12 months, as indicated by variceal bleeding, ascites, encephalopathy, Prothrombin or International Normalized Ratio (INR) prolonged to >1.7 x upper limit of normal (ULN), serum bilirubin > 2 mg/dl or albumin < 3.5 g/dl (i.e. Child-Pugh grade B, score > 7)
* For non-cirrhotic cohorts: Any previous liver biopsy consistent with cirrhosis. For cirrhotic cohorts: Any liver biopsy or fibroscan result from last 2 years excluding liver cirrhosis.
* Positive test for human immunodeficiency virus (HIV) or hepatitis B antigen at screening
* Current alcohol or drug abuse, or history of the same, within the past six (6) months. Exception: Occasional use of cannabis is not an exclusion criterion. The investigator must however instruct the patient that consumption of cannabis is not allowed during the treatment period.
* Any concurrent disease (cardiovascular, pulmonary, renal, haematological, neurological, psychiatric, immunologic, metabolic or endocrine dysfunction) if clinically significant based on the investigator's medical assessment at screening. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or may influence the results of the study or the patient's ability to participate in the study. Exclusion is also necessary for any pre-existing cardiac abnormality by history.
* Clinically significant abnormalities at screening ECG, including but not limited to a QTc longer than 435 msec, Pulse Rate > 240 msec at baseline and any bundle branch block pattern, but not necessarily non-specific T wave abnormalities
* History of malignancy (except for previously cured squamous cell or basal cell carcinoma)
* Patients treated with any interferon (IFN) (approved or investigational) or Peg-IFN and/or Ribavirin within 3 months prior to screening
* Planned or concurrent usage of any other pharmacological therapy including any antiviral therapy or vaccination from 7 days before treatment and during treatment
* Usage of any investigational drug within thirty (30) days prior to enrolment or 5 halflives, whichever is longer; or the planned usage of an investigational drug during the course of the current study
* Known hypersensitivity to drugs or excipients
* Patients with any one of the following laboratory values at screening:

  * Alanine transaminase (ALT) > 3x ULN, local lab
  * Aspartate aminotransferase (AST) > 3x ULN, local lab
  * Total bilirubin > 1.5x ULN, local lab, unless predominantly conjugated and reflecting Gilbert's disease
  * Alkaline phosphatase > 1.5x ULN, local lab
  * Prothrombin time (INR) > 1.5x ULN, central lab
  * Creatinine > 1x ULN, local lab
  * Urine protein / creatinine ratio > 0.3 g protein / g creatinine, central lab
  * Alpha-1-microglobulin / creatinine in urine > 1x ULN, central lab
  * Platelet count < 100,000 / mm3, central lab
  * White Blood cell count < 2000 cells/mm3, central lab
  * Absolute neutrophile count < 1500 cells, central lab
  * Hemoglobin < 12 g/dL, central lab
  * For patients with liver cirrhosis:

    * ALT > 5x ULN, local lab
    * AST > 5x ULN, local lab
    * Platelet count < 70,000 / mm3, central lab
* Patients with any clinically significant laboratory abnormalities based on the investigator's medical assessment at screening
* Positive urine test for drug abuse at screening
* Prior randomisation into this trial
* Inability to comply with the protocol
* Patients with ongoing or historical photosensitivity or recurrent rash
* Alpha fetoprotein value (AFP) > 100 ng/ml; if AFP is > 20 and ≤ 100 ng/ml, patients can be included if liver cancer is excluded by a current imaging study (i.e. ultrasound, computer tomography scan or magnetic resonance imaging)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: acronyms used in pre-assignment details: International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP)
Pre-assignment Details: Each patient participating in the trial (or the patient's legally accepted representative) provided written informed consent according to ICH GCP and the regulatory and legal requirements of the participating country. All subjects were informed that they were free to withdraw their consent at any time during the study without penalty or prejudice.
Groups:
- Placebo Fibrosis: Placebo (as tablet, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
- DBV 100mg Fibrosis: Deleobuvir (DBV) 100mg (as tablet, 2x 50mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
- DBV 200mg Fibrosis: DBV 200mg (as tablet, 1x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
- DBV 400mg Fibrosis: DBV 400mg (as tablet, 2x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
- DBV 400mg Cirrhosis: DBV 400mg (as tablet, 2x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with cirrhosis
- DBV 600mg Cirrhosis: DBV 600mg (as tablet, 3x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with cirrhosis
- DBV 800mg Fibrosis: DBV 800mg (as tablet, 4x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
- DBV 1200mg Fibrosis: DBV 1200mg (as tablet, 6x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
Period: Overall Study
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Started | 15 (15 subjects randomized, 14 subjects treated with at least one dose, 1 subject was not treated) | 9 | 9 | 9 | 8 | 6 (6 subjects randomized, 5 subjects treated with at least one dose, 1 subject was not treated) | 9 | 10
Completed | 14 | 9 | 9 | 8 | 7 | 5 | 8 | 10
Not Completed | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — not treated | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) included all patients who were dispensed study medication and were documented to have taken at least one dose of study treatment, regardless of randomisation. Full analysis set (FAS) included all randomised patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Groups:
- DBV 100mg Fibrosis: DBV 100mg (as tablet, 2x 50mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days in patients with fibrosis
- Total: Total of all reporting groups
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis | Total
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.1) | 50.3 (11.9) | 51.7 (8.5) | 52.3 (8.7) | 55.4 (7.0) | 56.2 (8.1) | 47.3 (12.7) | 46.8 (8.6) | 50.24 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 1 | 2 | 1 | 2 | 0 | 15
  Male | 9 | 8 | 6 | 8 | 6 | 4 | 7 | 10 | 58

OUTCOME MEASURES:

1. Primary Outcome: Virologic Response (VR)
Description: Virologic response was defined as a ≥ 1 log10 reduction in serum Hepatitis C virus (HCV) Ribonucleic acid (RNA) level from baseline at any time from the start of administration of treatment up to day 5. In this Outcome Measure the percentage of participants with virologic response is presented.
Time Frame: Baseline (Visit 2_2 at planned time 5 minutes prior to first administration of trial drug), up to day 5
Population: The full analysis set (FAS) included all randomised patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10
percentage of participants | 14.3 [4 to 40] | 22.2 [7 to 56] | 55.6 [26 to 81] | 88.9 [55 to 97] | 87.5 [52 to 97] | 100 [61 to 100] | 88.9 [55 to 97] | 100 [76 to 100]

2. Secondary Outcome: Time Dependent Change From Baseline in Viral Load (VL)
Description: Change of VL from baseline to day 7 is presented (VL at timepoint minus VL at baseline). Acronym used within the categories: planned time (PTM). The number of participants analysed displays the number of participants included in the analysis set whereas the number of participants for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Baseline, up to day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 (U/L)
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10
log10 (U/L)
  PTM 2:00 hours; N (per arm): 14/8/9/9/8/5/8/10 | -0.01 (0.15) | -0.03 (0.15) | -0.06 (0.26) | -0.13 (0.11) | 0.09 (0.10) | -0.01 (0.16) | 0.05 (0.25) | 0.03 (0.11)
  PTM 4:00 hours; N (per arm): 14/8/9/9/8/5/9/10 | -0.11 (0.09) | -0.02 (0.21) | -0.16 (0.18) | -0.25 (0.17) | -0.07 (0.22) | -0.03 (0.34) | -0.26 (0.17) | -0.15 (0.20)
  PTM 7:55 hours; N (per arm): 14/8/9/9/8/5/9/9 | -0.16 (0.37) | -0.33 (0.37) | -0.53 (0.60) | -0.96 (0.51) | -0.90 (0.53) | -1.05 (0.30) | -1.41 (0.53) | -1.11 (0.51)
  PTM 10:00 hours; N (per arm): 14/8/9/9/8/5/9/10 | -0.06 (0.19) | -0.55 (0.49) | -0.80 (0.59) | -1.21 (0.60) | -1.26 (0.53) | -1.57 (0.56) | -1.82 (0.59) | -1.59 (0.54)
  PTM 15:55 hours; N (per arm): 14/8/9/9/8/5/9/10 | -0.00 (0.19) | -0.53 (0.57) | -0.96 (0.78) | -1.66 (0.96) | -1.89 (0.69) | -2.30 (0.55) | -2.40 (0.76) | -2.31 (0.57)
  PTM 18:00 hours; N (per arm): 14/8/9/9/8/5/9/10 | -0.01 (0.18) | -0.43 (0.55) | -0.94 (0.69) | -1.64 (0.96) | -1.96 (0.69) | -2.49 (0.57) | -2.51 (0.86) | -2.40 (0.63)
  PTM 23:55 hours; N (per arm): 14/8/9/9/7/5/9/10 | 0.01 (0.17) | -0.53 (0.64) | -0.93 (0.82) | -1.67 (1.02) | -2.03 (0.79) | -2.75 (0.77) | -2.46 (1.04) | -2.45 (0.83)
  PTM 47:55 hours; N (per arm): 13/7/9/9/7/5/9/10 | -0.01 (0.18) | -0.46 (0.65) | -1.14 (1.26) | -1.79 (1.25) | -2.43 (0.88) | -3.14 (0.67) | -3.00 (1.14) | -3.01 (0.59)
  PTM 71:55 hours; N (per arm): 14/8/9/8/7/5/9/10 | -0.06 (0.16) | -0.50 (0.65) | -1.16 (0.92) | -1.84 (1.43) | -2.50 (0.93) | -3.17 (0.59) | -3.02 (1.30) | -2.97 (0.82)
  PTM 95:55 hours; N (per arm): 14/8/9/8/7/5/9/10 | -0.04 (0.27) | -0.61 (0.65) | -1.07 (0.94) | -1.87 (1.33) | -2.64 (1.19) | -3.19 (0.56) | -3.11 (1.23) | -2.94 (0.83)
  PTM 98:00 hours; N (per arm): 14/8/9/8/8/5/9/10 | -0.08 (0.26) | -0.66 (0.65) | -1.08 (0.89) | -1.93 (1.29) | -2.64 (1.13) | -3.13 (0.67) | -3.17 (1.29) | -3.01 (0.77)
  PTM 100:00 hours; N (per arm): 14/8/9/8/7/5/8/10 | -0.17 (0.24) | -0.60 (0.58) | -1.05 (0.80) | -1.94 (1.24) | -2.70 (1.23) | -3.16 (0.83) | -3.06 (1.40) | -3.02 (0.78)
  PTM 104:00 hours; N (per arm): 13/8/9/8/0/0/8/10 | -0.07 (0.19) | -0.77 (0.63) | -1.08 (0.92) | -1.96 (1.25) | NA (NA) — N=0 | NA (NA) — N=0 | -3.27 (1.30) | -3.11 (0.82)
  PTM 108:00 hours; N (per arm): 14/8/9/8/8/5/8/10 | -0.06 (0.20) | -0.56 (0.53) | -0.90 (1.01) | -1.80 (1.25) | -2.61 (1.17) | -3.19 (0.58) | -3.11 (1.20) | -3.03 (0.83)
  PTM 112:00 hours; N (per arm): 14/8/9/8/6/5/8/10 | -0.03 (0.18) | -0.56 (0.50) | -0.87 (0.85) | -1.64 (1.35) | -2.95 (1.25) | -3.12 (0.71) | -2.98 (1.30) | -2.91 (0.90)
  PTM 120:00 hours; N (per arm): 14/8/9/8/6/5/8/10 | -0.14 (0.50) | -0.37 (0.41) | -0.70 (0.68) | -1.47 (1.29) | -2.20 (1.46) | -2.97 (1.13) | -2.82 (1.40) | -2.64 (1.07)
  PTM 144:00 hours; N (per arm): 14/8/9/8/0/1/6/10 | 0.02 (0.76) | -0.19 (0.38) | -0.40 (0.93) | -0.76 (1.07) | NA (NA) — N=0 | -2.93 (NA) — N=1 | -1.88 (1.64) | -1.61 (0.87)

3. Secondary Outcome: Cmax
Description: Maximum measured concentration of Deleobuvir in plasma (Cmax) determined after the first dose.
Time Frame: 5 minutes (min) prior to the first dose of study medication and 30 minutes and 1:00, 2:00, 3:00, 4:00, 6:00, 7:55, 10:00, 12:00, 15:55, 18:00 hours (h) thereafter on day 1
Population: The PK set (PKS) included all patients in the full analysis set (FAS) with evaluable PK data. FAS included all randomised patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/millilitre (ng/mL)
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 5 | 9 | 10
nanogram/millilitre (ng/mL) | 320 (75.0) | 656 (73.1) | 3500 (22.1) | 4060 (70.1) | 6760 (50.6) | 5730 (74.4) | 9570 (35.9)

4. Secondary Outcome: Cmin
Description: Measured concentration of Deleobuvir in plasma determined immediately before the second dose (Cmin). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 8 | 8 | 9 | 8 | 5 | 9 | 10
ng/mL | 105 (83.1) | 210 (80.6) | 1190 (39.3) | 1520 (77.0) | 3470 (37.7) | 1800 (65.8) | 5090 (59.5)

5. Secondary Outcome: Tmax
Description: Time from dosing to maximum measured concentration (tmax) of Deleobuvir determined after the first dose.
Time Frame: as for outcome 3
Population: PKS
Measure: Median (Full Range); unit: hours (h)
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 5 | 9 | 10
hours (h) | 3.00 [2.00 to 4.17] | 3.03 [2.03 to 4.00] | 3.00 [2.00 to 4.00] | 4.00 [2.00 to 6.00] | 6.00 [4.00 to 6.00] | 4.00 [2.83 to 6.00] | 6.00 [4.00 to 6.00]

6. Secondary Outcome: AUC0-τ
Description: Area under the concentration-time curve of Deleobuvir in plasma over the interval 0 hour (h) to the next dose of trial medication (AUC0-τ) measured after first administration of trial drug.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hours/millilitre (ng*h/mL)
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 5 | 9 | 10
Nanogram*hours/millilitre (ng*h/mL) | 1410 (77.9) | 2820 (66.6) | 15900 (27.3) | 18600 (62.7) | 29500 (49.4) | 23600 (69.5) | 42400 (42.2)

7. Secondary Outcome: Cmax,ss
Description: The maximum measured concentration of Deleobuvir in plasma at steady state after the last dose of study drug (Cmax,ss).
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only)
Time Frame: 5 min prior to the first dose of study medication of Day 5; 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00, 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h thereafter
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 8 | 10
ng/mL | 391 (67.8) | 910 (80.3) | 3780 (46.3) | 6780 (76.7) | 15400 (80.4) | 9030 (103.0) | 16500 (66.7)

8. Secondary Outcome: Cmin,ss
Description: The minimum measured concentration of Deleobuvir in plasma at steady state (Cmin,ss).
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 7 | 10
ng/mL | 109 (98.5) | 201 (90.9) | 1150 (65.9) | 2340 (110.0) | 6920 (93.9) | 2100 (247.0) | 6630 (118.0)

9. Secondary Outcome: Tmax,ss
Description: Time from dosing to the maximum measured concentration of Deleobuvir at steady state after the last dose of study drug (tmax,ss) more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only)
Time Frame: as for outcome 7
Population: PKS
Measure: Median (Full Range); unit: h
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 8 | 10
h | 2.02 [1.00 to 4.00] | 4.00 [1.00 to 6.00] | 2.52 [1.00 to 4.00] | 4.00 [1.03 to 4.02] | 4.00 [0.50 to 4.00] | 4.00 [2.00 to 4.00] | 4.10 [1.00 to 6.30]

10. Secondary Outcome: AUCτ,ss
Description: Area under the concentration-time curve of Deleobuvir in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) measured after last dose of trial drug.
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 8 | 10
ng*h/mL | 1930 (79.0) | 4130 (79.1) | 17900 (37.1) | 36800 (82.7) | 86400 (78.1) | 43500 (118.0) | 88500 (83.3)

11. Secondary Outcome: AUC0-∞,ss
Description: Area under the concentration-time curve of Deleobuvir in plasma over the interval 0 hour (h) extrapolated to infinity at steady state (AUC0-∞,ss) measured after last administration of trial drug.
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 4 | 7 | 10
ng*h/mL | 2560 (91.8) | 5420 (87.6) | 22800 (41.6) | 54300 (110.0) | 153000 (108.0) | 51700 (159.0) | 129000 (119.0)

12. Secondary Outcome: λz,ss
Description: Terminal rate of Deleobuvir constant in plasma at steady state (λz,ss) measured after last dose of study drug.
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Median (Full Range); unit: 1/h
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 7 | 10
1/h | 0.189 [0.0976 to 0.264] | 0.180 [0.111 to 0.322] | 0.131 [0.110 to 0.186] | 0.117 [0.0869 to 0.209] | 0.117 [0.110 to 0.124] | 0.155 [0.115 to 0.273] | 0.145 [0.118 to 0.163]

13. Secondary Outcome: t1/2,ss
Description: Terminal half-life of Deleobuvir in plasma at steady state (t1/2,ss) measured after the last dose of study drug.
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Median (Full Range); unit: h
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 7 | 10
h | 3.67 [2.63 to 7.10] | 3.84 [2.15 to 6.24] | 5.31 [3.73 to 6.33] | 5.90 [3.32 to 7.98] | 5.95 [5.59 to 6.28] | 4.48 [2.54 to 6.02] | 4.79 [4.24 to 5.85]

14. Secondary Outcome: CL/F,ss
Description: Apparent clearance of Deleobuvir in plasma after oral administration at steady state (CL/F,ss) measured after the last dose of study drug.
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Millilitre per minute (mL/min)
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 7 | 10
Millilitre per minute (mL/min) | 865 (79.0) | 806 (79.1) | 372 (37.1) | 181 (82.7) | 116 (78.1) | 319 (132.0) | 226 (83.3)

15. Secondary Outcome: Vz/F,ss
Description: Apparent volume of Deleobuvir distribution during the terminal phase λz following an oral dose at steady state (Vz/F,ss) after the last dose of study drug.
  more detailed time frame information: 5 minutes (min) prior to the first dose of study medication of Day 5 (-0:05) and 0:30, 1:00, 2:00, 3:00*, 4:00, 6:00, 8:00*, 10:00, 12:00, 16:00, 24:00, 48:00 h thereafter; Assigned to the planned time points 95:55, 96:30, 97:00, 98:00 99:00*, 100:00, 102:00, 104:00*, 106:00, 108:00, 112:00, 120:00, 144:00 h (*At these time points, in patients with cirrhosis only). The number of participants analysed displays the number of participants with available data at the timepoints of interest.
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (L)
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 8 | 7 | 5 | 7 | 10
Litre (L) | 279 (53.1) | 254 (49.8) | 164 (41.4) | 83.9 (58.2) | 59.7 (72.8) | 110 (108.0) | 96.8 (86.5)

16. Secondary Outcome: Plasma Concentration Time Profiles
Description: Individual drug plasma concentrations of Deleobuvir after multiple oral administration. Within the categories PTM means planned time. The number of participants analysed displays the number of participants included in the analysis data set whereas the number of participants for each timepoint displays the number of participants with available data at that timepoint. Below the limit of quantification (BLQ) is abbreviated.
Time Frame: up to day 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 5 | 9 | 10
ng/mL
  PTM 0.5 hours; N(per Arm)=6/6/7/8/3/5/9) | 54.6 (328.0) | 15.1 (57.7) | 163 (214.0) | 45.4 (632.0) | NA (NA) — 2 of 5 samples BLQ, no descriptive statistics calculated | NA (NA) — 4 of 9 samples BLQ, no descriptive statistics calculated | 124 (1250.0)
  PTM 1 hour; N(per Arm)=7/9/9/8/5/8/10) | 91.4 (111.0) | 53.0 (387.0) | 427 (569.0) | 597 (168.0) | 177 (258.0) | 519 (570.0) | 647 (275.0)
  PTM 2 hours; N(per Arm)=9/9/9/8/5/9/10) | 208 (199.0) | 246 (133.0) | 2290 (70.8) | 1720 (62.4) | 1390 (112.0) | 1650 (240.0) | 1780 (208.0)
  PTM 3 hours; N(per Arm)=9/9/9/8/5/9/10) | 162 (213.0) | 476 (74.9) | 2830 (41.8) | 2950 (50.1) | 3330 (89.9) | 3750 (106.0) | 4330 (110.0)
  PTM 4 hours; N(per Arm)=9/9/9/8/5/9/10) | 274 (70.0) | 574 (73.8) | 2800 (35.6) | 3740 (70.4) | 5060 (83.2) | 4920 (78.0) | 6930 (64.9)
  PTM 6 hours; N(per Arm)=9/8/9/8/5/9/10) | 181 (69.5) | 377 (57.6) | 2030 (42.9) | 2760 (89.7) | 6250 (57.4) | 3350 (75.0) | 8890 (34.6)
  PTM 7.917 hours; N(per Arm)=8/8/9/8/5/9/10) | 105 (83.1) | 210 (80.6) | 1190 (39.3) | 1520 (77.0) | 3470 (37.7) | 1800 (65.8) | 5090 (59.5)
  PTM 10 hours; N(per Arm)=9/9/9/8/5/9/10) | 282 (88.7) | 646 (170.0) | 4170 (93.7) | 2580 (79.7) | 5770 (88.6) | 4120 (75.4) | 9720 (48.9)
  PTM 12 hours; N(per Arm)=9/9/9/8/5/9/10) | 161 (66.2) | 769 (92.8) | 3300 (31.5) | 3500 (74.8) | 7340 (49.6) | 7290 (48.2) | 12700 (68.1)
  PTM 15.917 hours; N(per Arm)=9/9/9/7/5/9/10) | 73.7 (101.0) | 222 (90.5) | 1180 (32.7) | 1600 (76.1) | 5230 (49.2) | 2220 (96.1) | 5120 (112.0)
  PTM 18 hours; N(per Arm)=9/9/9/8/5/9/10) | 265 (69.7) | 379 (155.0) | 2520 (82.6) | 2870 (97.5) | 5340 (67.9) | 3060 (165.0) | 8100 (108.0)
  PTM 23.917 hours; N(per Arm)=9/9/9/7/5/9/10) | 164 (98.1) | 531 (78.1) | 2290 (48.8) | 3570 (113.0) | 7690 (61.5) | 4840 (91.4) | 13800 (64.8)
  PTM 47.917 hours; N(per Arm)=9/9/9/7/5/9/10) | 154 (81.4) | 403 (96.6) | 2200 (32.6) | 3490 (119.0) | 9200 (83.6) | 4680 (157.0) | 12000 (89.1)
  PTM 71.917 hours; N(per Arm)=9/9/8/7/5/9/10) | 164 (98.0) | 378 (70.7) | 1670 (40.6) | 3420 (90.0) | 11500 (77.2) | 3170 (219.0) | 9440 (202.0)
  PTM 95.917 hours; N(per Arm)=9/9/8/7/5/9/10) | 158 (93.7) | 383 (88.7) | 1880 (34.0) | 2820 (86.8) | 5600 (192.0) | 3120 (224.0) | 7820 (133.0)
  PTM 96.5 hours; N(per Arm)=9/9/8/7/5/9/10) | 149 (90.6) | 366 (84.7) | 1830 (51.1) | 3220 (85.0) | 8360 (92.7) | 3330 (181.0) | 7840 (114.0)
  PTM 97 hours; N(per Arm)=9/9/8/7/5/9/9) | 209 (88.4) | 427 (86.0) | 2400 (56.7) | 3610 (76.3) | 8510 (73.9) | 4350 (142.0) | 9460 (118.0)
  PTM 98 hours; N(per Arm)=9/9/8/7/5/9/10) | 313 (64.3) | 503 (105.0) | 2760 (49.7) | 4620 (77.0) | 10000 (74.3) | 7390 (118.0) | 11400 (86.7)
  PTM 99 hours; N(per Arm)=9/9/8/7/5/8/10) | 300 (70.4) | 565 (108.0) | 2820 (37.2) | 5120 (93.5) | 11200 (79.5) | 7990 (94.2) | 12200 (72.9)
  PTM 100 hours; N(per Arm)=9/9/8/7/5/8/10) | 329 (86.9) | 658 (109.0) | 2790 (50.2) | 6210 (89.9) | 14800 (86.7) | 7740 (107.0) | 14000 (74.7)
  PTM 102 hours; N(per Arm)=9/9/8/7/5/8/10) | 199 (92.7) | 492 (99.4) | 1630 (70.6) | 4600 (102.0) | 11400 (76.6) | 4450 (144.0) | 11200 (91.6)
  PTM 104 hours; N(per Arm)=9/9/8/7/5/7/10) | 124 (113.0) | 254 (109.0) | 867 (73.1) | 2710 (119.0) | 7450 (91.5) | 2230 (222.0) | 6830 (150.0)
  PTM 106 hours; N(per Arm)=9/9/8/7/5/7/10) | 76.2 (121.0) | 158 (115.0) | 553 (74.8) | 1720 (153.0) | 5260 (115.0) | 1200 (316.0) | 4370 (190.0)
  PTM 108 hours; N(per Arm)=9/9/8/7/5/7/10) | 52.5 (136.0) | 92.7 (136.0) | 321 (79.0) | 1160 (171.0) | 4040 (120.0) | 681 (403.0) | 2780 (314.0)
  PTM 112 hours; N(per Arm)=9/9/8/7/5/7/10) | 20.8 (138.0) | 39.9 (157.0) | 153 (82.6) | 553 (211.0) | 1890 (130.0) | 239 (436.0) | 1110 (444.0)
  PTM 120 hours; N(per Arm)= 5/6/8/ 7/5/7/10) | NA (NA) — 4 of 9 samples below limit of quantification (BLQ). 5 values were reportable (5 of 9 = total N of 55.6%), no descriptive statistics calculated. A total N of 66.7 % (2/3) of reportable values is needed. | 20.2 (126.0) | 59.0 (75.9) | 219 (269.0) | 699 (185.0) | 67.2 (384.0) | 316 (512.0)
  PTM 144 hours; N(per Arm)= 1/1/5/ 5/5/4/10) | NA (NA) — 8 of 9 samples BLQ, no descriptive statistics calculated | NA (NA) — 8 of 9 samples BLQ, no descriptive statistics calculated | NA (NA) — 3 of 9 samples BLQ. Another subject did not have PK sampling past 48 hours. 5 values were reportable (5 of 9 = total N of 55.6%), no descriptive statistics calculated. A total N of 66.7 % (2/3) of reportable values is needed. | 36.2 (272.0) | 56.2 (186.0) | NA (NA) — 3 of 9 samples BLQ and another sample excluded, no descriptive statistics calculated | 20.1 (175.0)

17. Secondary Outcome: Number of Patients With Clinically Significant Changes in Vital Signs (Pulse Rate, Systolic and Diastolic Blood Pressure).
Description: Number of patients with clinically significant changes in vital signs (pulse rate, systolic and diastolic blood pressure) presents the number of patients with an reported adverse event which has a symptom in changes in vital signs. Vascular disorders was identified as changes in vital signs. The number of participant with vascular disorders is presented in this outcome measure
Time Frame: Baseline, up to day 14
Population: The treated set (TS) included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment, regardless of randomisation.
Measure: Number; unit: participants
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10
participants | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Patients With Abnormal Findings in 12-lead ECG (Electrocardiogram)
Description: Number of patients with a new onset of an abnormal finding by central assessment are presented.
Time Frame: up to 14 days
Population: Treated set (TS) included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment, regardless of randomisation. Only patients included having no missing ECG measurements .
Measure: Number; unit: participants
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 16 | 5 | 9 | 9
participants
  None | 13 | 9 | 9 | 12 | 5 | 8 | 7
  Sinus rhythm | 1 | 0 | 0 | 3 | 0 | 1 | 2
  Conduction | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Morphology | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myocardial infarction | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ST segment | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T-wave | 0 | 0 | 0 | 0 | 0 | 0 | 0
  U-wave | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Patients With Abnormal Changes in Laboratory Tests
Description: Number of patients with abnormal changes in safety laboratory tests including urine protein diagnostics, and adrenocorticotropic hormone (ACTH) and cortisol measurements resulted in adverse events.
Time Frame: Baseline, up to day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Patients With Adverse Events
Description: Number of patients with any adverse event (AE)
Time Frame: up to 14 days
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10
participants | 4 | 2 | 3 | 7 | 5 | 4 | 6 | 9

21. Secondary Outcome: Number of Patients With Abnormal Findings in Physical Examination
Description: The number of patients with abnormal findings in physical examination presents the number of patients with any treatment-emergent adverse events in this study.
Time Frame: up to day 14
Population: as for outcome 17
Measure: Number; unit: participants
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 9 | 8 | 5 | 9 | 10
participants | 4 | 2 | 3 | 7 | 5 | 4 | 6 | 9

22. Secondary Outcome: Assessment of Global Tolerability on a 4-point Scale
Description: The global tolerability was presented on a four item scale: good, satisfactory, not satisfactory and bad. Rating was done by the investigator.
Time Frame: day 6
Population: as for outcome 17
Measure: Number; unit: participants
Groups:
- DBV 400mg: DBV 400mg (as tablet, 2x 200mg, oral) administered 3 times (every 8 hours) daily after a meal for 5 days. Subgroup of patients in fibrosis and in cirrhosis presented in one arm.
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 17 | 5 | 9 | 10
participants
  Good | 11 | 9 | 8 | 12 | 4 | 8 | 9
  Satisfactory | 3 | 0 | 1 | 3 | 1 | 0 | 1
  Not satisfactory | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Bad | 0 | 0 | 0 | 0 | 0 | 1 | 0

23. Secondary Outcome: Body Temperature
Description: The body temperature will be presented as the mean values in visit 1 and visit 7. The number of participants analysed displays the number of participants included in the analysis set whereas the numbers for each timepoint display the number of participants with available data at that timepoint.
Time Frame: Visit 1, Visit 7
Population: Treated set.
Measure: Mean (Standard Deviation); unit: degree (°C)
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Number analyzed (Participants) | 14 | 9 | 9 | 17 | 5 | 9 | 10
degree (°C)
  Visit 1 (N=7/5/8/14/5/7/6) | 36.429 (0.287) | 36.780 (0.455) | 36.513 (0.557) | 36.550 (0.641) | 35.760 (0.709) | 36.686 (0.248) | 36.517 (0.567)
  Visit 7 (N=13/9/9/15/5/8/10) | 36.400 (0.283) | 36.656 (0.403) | 36.156 (0.265) | 36.307 (0.451) | 35.540 (0.445) | 36.125 (0.287) | 36.320 (0.744)

ADVERSE EVENTS:
Time Frame: Assessment of adverse events from the baseline up to 14 days
Description: The treated set (TS) included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment, regardless of randomisation.
Arm/Group | Placebo Fibrosis | DBV 100mg Fibrosis | DBV 200mg Fibrosis | DBV 400mg Fibrosis | DBV 400mg Cirrhosis | DBV 600mg Cirrhosis | DBV 800mg Fibrosis | DBV 1200mg Fibrosis
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9 | 0/9 | 0/9 | 0/8 | 0/5 | 1/9 | 0/10
Other Adverse Events (participants affected / at risk) | 4/14 | 2/9 | 3/9 | 7/9 | 5/8 | 4/5 | 6/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Fibrosis (N=14) | DBV 100mg Fibrosis (N=9) | DBV 200mg Fibrosis (N=9) | DBV 400mg Fibrosis (N=9) | DBV 400mg Cirrhosis (N=8) | DBV 600mg Cirrhosis (N=5) | DBV 800mg Fibrosis (N=9) | DBV 1200mg Fibrosis (N=10)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Fibrosis (N=14) | DBV 100mg Fibrosis (N=9) | DBV 200mg Fibrosis (N=9) | DBV 400mg Fibrosis (N=9) | DBV 400mg Cirrhosis (N=8) | DBV 600mg Cirrhosis (N=5) | DBV 800mg Fibrosis (N=9) | DBV 1200mg Fibrosis (N=10)
Cardiovascular disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 7
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Irritability (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urine colour abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 0 | 0 | 1 | 2 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.